CLINICAL TRIAL: NCT00461032
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Parallel Group 8-week Study to Evaluate the Efficacy and Safety of Chewable Montelukast When Initiated at the Start of the School Year in Pediatric Patients With Chronic Asthma
Brief Title: Montelukast Back to School Asthma Study (0476-340)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-340; MK0476-340; 2007_539
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): montelukast
  Interventions: Drug: montelukast
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: montelukast — montelukast 5 mg tablet Once a day (QD) for 8 weeks
  Arms: 1
Drug: Comparator: Placebo — Placebo to montelukast QD for 8 weeks
  Arms: 2

SUMMARY:
This study, in children with chronic asthma, evaluates the number of days of worsening asthma during 8 weeks of treatment with montelukast after treatment is started for the first day of school.

ELIGIBILITY:
Inclusion Criteria:

* Male and female non-smoking Participants, ages 6 to 14 years, with chronic asthma, history of at least one asthma exacerbation associated with a cold within the past year and a documented history of asthma that required treatment with any asthma medication within 6 months prior to Visit 1

Exclusion Criteria:

* Participant cannot have any other acute or chronic pulmonary disorder, or hospitalization for asthma more than three times within one year prior to signing informed consent

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1162 (Actual)
Dates: Start 2006-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Weiss KB, Gern JE, Johnston NW, Sears MR, Jones CA, Jia G, Watkins MW, Smugar SS, Edelman JM, Grant EN. The Back to School asthma study: the effect of montelukast on asthma burden when initiated prophylactically at the start of the school year. Ann Allergy Asthma Immunol. 2010 Aug;105(2):174-81. doi: 10.1016/j.anai.2010.04.018. Epub 2010 Jul 1. PMID 20674830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 165 sites in the US and Canada.
  Therapy period: June to November 2006 (including screening period).
Pre-assignment Details: Participants who were hospitalized for asthma in the 4 weeks prior to randomization or who required excluded medications were excluded from randomization.
Groups:
- Placebo: Montelukast matching-image placebo tablet taken orally once daily at bedtime for 8 weeks.
- Montelukast 5 mg: Montelukast 5 mg chewable tablet taken orally once daily (OD) at bedtime for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Montelukast 5 mg
Started | 582 | 580
Completed | 545 | 536
Not Completed | 37 | 44
Not completed — Adverse Event | 5 | 6
Not completed — Lack of Efficacy | 5 | 1
Not completed — Lost to Follow-up | 7 | 12
Not completed — Protocol Violation | 4 | 4
Not completed — Withdrawal by Subject | 7 | 15
Not completed — Patient Moved or Relocated | 2 | 1
Not completed — Other | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast 5 mg | Total
Number analyzed (Participants) | 582 | 580 | 1162
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (2.5) | 9.9 (2.4) | 9.9 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 225 | 461
  Male | 346 | 355 | 701
Daytime Asthma Symptom Score [Mean (Standard Deviation); unit: Units on a Scale] — The Participant or parent/guardian scored his/her/child's symptoms [from 0 (best) to 5 (worst)] on a daily basis. Scores were entered into a Participant diary during the 2-week period prior to the start of the study drug.
  Units on a Scale | 1.32 (1.81) | 1.35 (1.94) | 1.34 (1.88)
β-Agonist Use [Mean (Standard Deviation); unit: puffs/day] — The number of puffs used per day was entered by the Participant or parent/guardian into a Participant diary during the 2-week period prior to the start of the study drug.
  puffs/day | 0.62 (1.11) | 0.54 (0.94) | 0.58 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Days With Worsening Asthma (as Measured on Daily Diaries) in Pediatric Asthmatic Participants
Description: A day of worsening asthma is a day with: increase from baseline in β-agonist use (> 70% and a min increase of 2 puffs); > 50% increase from baseline in daytime symptoms score; awake "all night"; increase from baseline in inhaled corticosteroid use ≥ 100% or oral corticosteroid rescue for worsening asthma; or unanticipated healthcare utilization.
Time Frame: 8 Week treatment period initiated at the beginning of a school year
Population: The primary efficacy analysis was based on full-analysis-set (FAS) population. This included all randomized participants who received at least one dose of double-blinded therapy and had a valid efficacy measurement. The percent of worsening asthma days was calculated from at least 7 days of diary data. Missing diary data were not imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Days
Arm/Group | Placebo | Montelukast 5 mg
Number analyzed (Participants) | 499 | 499
Percentage of Days | 27.23 [24.25 to 30.00] | 24.26 [21.52 to 27.01]

2. Secondary Outcome: Number of Participants With the Occurrence of One or More Health Care Utilizations (as Measured on Daily Diaries)
Description: Health care utilization is defined as unanticipated asthma care in an office or clinic, emergent or hospital setting.
Time Frame: 8 Week treatment period initiated at the beginning of a school year
Population: The analysis was based on the FAS population. This included all randomized participants who received at least 1 dose of study medication and had a valid efficacy measurement. Occurrence of one or more health care utilization was derived from the available diary data and was set to missing if no diary data were available.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast 5 mg
Number analyzed (Participants) | 476 | 466
Participants
  Participants requiring Health Care Utilization | 70 | 55
  Participants not requiring Health Care Utilization | 406 | 411

3. Secondary Outcome: Percentage of Days With Increased β-agonist Use by >70% and a Minimum Increase of 2 Puffs From Baseline (as Measured on Daily Diaries) in Pediatric Asthmatic Participants
Time Frame: 8 Week treatment period initiated at the beginning of a school year
Population: The secondary efficacy analysis was based on full-analysis-set (FAS) population. This included all randomized participants who received at least one dose of double-blinded therapy and had valid efficacy measurement for at least 7 days of diary data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Days
Arm/Group | Placebo | Montelukast 5 mg
Number analyzed (Participants) | 491 | 495
Percentage of Days | 7.02 [5.80 to 8.23] | 6.04 [4.84 to 7.24]

4. Secondary Outcome: Percentage of Days With Increased Daytime Asthma Symptom Score by >50% From Baseline (as Measured on Daily Diaries) in Pediatric Asthmatic Participants
Description: Daytime asthma symptom score was calculated as the sum of the responses (0 (best) to 5 (worst)) to three daytime symptom questions.
Time Frame: 8 Week treatment period initiated at the beginning of a school year
Population: The secondary efficacy analysis was based on full-analysis-set (FAS) population. This included all randomized participants who received at least one dose of double-blinded therapy and had a valid efficacy measurement. Variables that were measured as the average over the treatment period were defined from at least 7 days of evaluable diary data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Days
Arm/Group | Placebo | Montelukast 5 mg
Number analyzed (Participants) | 491 | 496
Percentage of Days | 17.4 [15.33 to 19.47] | 16.03 [13.99 to 18.07]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected during the 8 week, double-blind treatment period, and up to and including 14 days after the last dose of study therapy
Description: The number of participants listed in the AE tables (566 placebo & 566 montelukast) is the number that received treatment. 16 placebo & 14 montelukast randomized participants did not receive treatment.
  Although a participant may have 2 or more AEs they are counted only once in a category. The same participant may appear in other categories.
Arm/Group | Placebo | Montelukast 5 mg
Serious Adverse Events (participants affected / at risk) | 1/566 | 4/566
Other Adverse Events (participants affected / at risk) | 189/566 | 191/566
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=566) | Montelukast 5 mg (N=566)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=566) | Montelukast 5 mg (N=566)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphangioma (Congenital, familial and genetic disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 3
Conjunctivitis (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Stomach discomfort (Gastrointestinal disorders) | 1 | 3
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 5
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 3
Pyrexia (General disorders) | 5 | 9
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Acarodermatitis (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 4 | 3
Body tinea (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 6 | 2
Bronchitis acute (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 2 | 0
Eye infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 6 | 8
Herpes simplex (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 3
Impetigo (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 24 | 31
Otitis externa (Infections and infestations) | 3 | 0
Otitis media (Infections and infestations) | 3 | 7
Otitis media acute (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 2
Pharyngitis streptococcal (Infections and infestations) | 7 | 9
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 11 | 15
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 45 | 31
Urinary tract infection (Infections and infestations) | 1 | 1
Varicella (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 10 | 5
Viral upper respiratory tract infection (Infections and infestations) | 11 | 7
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 7 | 8
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 3 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Mood swings (Psychiatric disorders) | 0 | 1
Sleep terror (Psychiatric disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 1
Nipple swelling (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 28 | 21
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 4
Endodontic procedure (Surgical and medical procedures) | 0 | 1
Wisdom teeth removal (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.